CLINICAL TRIAL: NCT00731640
Title: Clinical Outcomes With AcrySof ReSTOR Aspheric Apodized Diffractive Intraocular Lens (IOL) in One Eye and a Contralateral Monofocal IOL or Phakic Eye
Brief Title: Contralateral ReSTOR / Monofocal or Phakic Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Rick Potvin/Director - Global Scientific Market Affairs, Alcon Research
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M07-012
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2010-03-16 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2010-03

CONDITIONS: Cataracts
Keywords: AcrySof; ReSTOR; Multifocal; Intraocular Lens
MeSH Terms: conditions — Cataract

ARMS (2):
- Monofocal (Active Comparator): Patients unilaterally implanted with ReSTOR lens in one eye and previously implanted with monofocal Intraocular lens (IOL) (unspecified) in other eye
  Interventions: Device: ReSTOR
- Phakic (Active Comparator): Patients unilaterally implanted with ReSTOR lens in one eye and phakic in the other eye with no necessary cataract removal impending
  Interventions: Device: ReSTOR

INTERVENTIONS:
Device: ReSTOR — AcrySof ReSTOR +4 Intraocular Lens (IOL) unilaterally implanted

SUMMARY:
Bilateral evaluation of unilateral implantation of ReSTOR and contralateral monofocal or phakic eye.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral operable cataract
* Candidate for presbyopic intraocular lens (IOL)

Exclusion Criteria:

* Ocular comorbidities compromising primary outcome
* Bilateral cataracts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a retrospective study that required patients with unilateral implantation of the AcrySof ReSTOR Intraocular Lens (IOL). Patients were to be free of conditions or ocular co-morbidities that may affect visual acuity.
Pre-assignment Details: During the preoperative exam, subjects were examined to ensure they met the inclusion/exclusion criteria. Only subjects who signed an informed consent and qualified to be in the study by meeting all inclusion/exclusion criteria were enrolled. This study was not randomized.
Period: Overall Study
Arm/Group | Monofocal | Phakic
Started | 20 | 32
Completed | 20 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monofocal | Phakic | Total
Number analyzed (Participants) | 20 | 32 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 23 | 31
  >=65 years | 12 | 9 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 11 | 19 | 30

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Uncorrected Visual Acuity (VA) is measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better visual acuity.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Monofocal | Phakic
Number analyzed (Participants) | 20 | 32
LogMar
  Distance | -0.04 (0.09) | -0.01 (0.09)
  Intermediate | 0.14 (0.13) | 0.18 (0.15)
  Near (Preferred Distance) | 0.04 (0.10) | 0.09 (0.12)

2. Secondary Outcome: Contrast Sensitivity
Description: Contrast sensitivity is the measurement of one's ability to detect slight changes in luminance before it becomes indistinguishable. It is measured in logarithmic (log) units by means of an illuminated box, the CSV 1000 by Vector Vision. A higher value for the logarithmic units translates to better contrast sensitivity.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Log Units
Arm/Group | Monofocal | Phakic
Number analyzed (Participants) | 20 | 32
Log Units
  Photopic CS, 3 cycles per degree (cpd) | 1.95 (0.13) | 1.90 (0.13)
  Mesopic CS, 3 cpd | 1.85 (0.18) | 1.84 (0.19)
  Mesopic w/Glare CS, 3 cpd | 1.82 (0.18) | 1.81 (0.22)
  Photopic CS, 6 cpd | 2.10 (0.24) | 2.05 (0.20)
  Mesopic CS, 6 cpd | 1.76 (0.36) | 1.62 (0.39)
  Mesopic w/Glare CS, 6 cpd | 1.73 (0.23) | 1.57 (0.56)
  Photopic CS, 12 cpd | 1.78 (0.26) | 1.66 (0.27)
  Mesopic CS, 12 cpd | 1.18 (0.51) | 0.95 (0.51)
  Mesopic w/Glare CS, 12 cpd | 1.21 (0.38) | 0.88 (0.54)
  Photopic CS, 18 cpd | 1.18 (0.39) | 1.14 (0.31)
  Mesopic CS, 18 cpd | 0.61 (0.52) | 0.49 (0.58)
  Mesopic w/Glare CS, 18 cpd | 0.57 (0.41) | 0.40 (0.52)

3. Secondary Outcome: Patient Satisfaction
Description: Average rating of patient satisfaction based on a patient survey. The survey had a 10 point scale (10 being most satisfied and 0 being most unsatisfied).
Time Frame: 6 Months Postoperative
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Monofocal | Phakic
Number analyzed (Participants) | 20 | 32
Units on a Scale | 6.85 (2.41) | 7.63 (2.24)

4. Secondary Outcome: Spectacle Independence
Description: The percentage of patients reporting spectacle independence (no longer needing to wear glasses).
Time Frame: 6 Months
Measure: Number; unit: Percentage of Participants
Arm/Group | Monofocal | Phakic
Number analyzed (Participants) | 20 | 32
Percentage of Participants | 65 | 56

ADVERSE EVENTS:
Arm/Group | Monofocal | Phakic
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/32
Other Adverse Events (participants affected / at risk) | 0/20 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Specify: No paper that incorporates Sponsor Confidential Information will be submitted for publication without Sponsor's prior written agreement.